CLINICAL TRIAL: NCT01244412
Title: Assessment of Prototype Hand-held Fundus Camera
Status: Terminated | Type: Observational
Why Stopped: The PI wanted to make additional changes to the hand held camera therefore he terminated the study rather than continue with an outdated camera design.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, david kleinman, Medical Doctor, University of Rochester
Other Study IDs: LUM-001
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Evaluate Performance of New Fundus Camera
Keywords: Fundus photography

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
This is the proof of concept study to evaluate the performance of an early stage prototype of a hand-held fundus camera.

DETAILED DESCRIPTION:
We tested a novel fundus camera. The images obtained were acceptable to move to the next step in development.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 21 years of age
* Ability to give informed consent
* Willingness to spend up to 2 hours for photos
* 5 patients presumed to be normal
* 5 patients with abnormalities of the posterior pole of the retina or the optic nerve will be studied

Exclusion Criteria:

* Any known pathology felt by the Principal Investigator to be significant so as to preclude participation as a normal subject
* Monocular subjects
* Potential subjects may be excluded based on the Principal Investigator's judgement that they are not good subjects to photograph
* Children and vulnerable subjects will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Flaum Eye Institute-University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Imaged Subjects: Subjects imaged with hand held device
Period: Overall Study
Arm/Group | Imaged Subjects
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imaged Subjects
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1
Acceptability of Hand Held Fundus Photograph in comparison to traditional photgraph [Number; unit: participants] — Scale Image scored as follows
  1. Unacceptable: cannot see fundus detail
  2. Unacceptable: fundus detail visualized, but inadequate for meaningful analysis
  3. Acceptable: fundus detail visualized to make general comments, modest improvement image would be of sufficient quality for use
  4. Good: fundus detail visualized, meaningful analysis possible, std photo superior
  5. Excellent: fundus detail visualized as well as std photo
  6. Superior: fundus detail of higher quality than std photo
  Report number of participants with score of 3 or higher
  participants | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have an Acceptable Image (Image Score of 3 or Higher) of Their Eye With the Hand Held Camera
Description: Will determine if the hand held camera is comparable to the traditional table mount camera in quality of images. The quality of the image of the participant's eye taken with the hand held camera will be compared to the quality of the image taken with the table mount camera using the following scale. We will determine the number of participants who have a score of 3 or higher.
  Scale Image scored as follows
  1. Unacceptable: cannot see fundus detail
  2. Unacceptable: fundus detail visualized, but inadequate for meaningful analysis
  3. Acceptable: fundus detail visualized to make general comments, modest improvement image would be of sufficient quality for use
  4. Good: fundus detail visualized, meaningful analysis possible, std photo superior
  5. Excellent: fundus detail visualized as well as std photo
  6. Superior: fundus detail of higher quality than std photo
Time Frame: estimated 3 months
Measure: Number; unit: participants
Arm/Group | Imaged Subjects
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Arm/Group | Imaged Subjects
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
It was determined that the project should stop in order for more technical changes to be made on the prototype

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less